CLINICAL TRIAL: NCT02451306
Title: Cognitive Control and Functional Connectivity During Resting State in Patients With Heightened Risk of Bipolar Disorder - a Quetiapine Challenge
Brief Title: Effect of Quetiapine on Brain Activity Patterns in Patients With Heightened Risk of Bipolar Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: EK018/15
Record Dates: First submitted 2015-04-22; First posted 2015-05-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Depression; Bipolar Disorder
MeSH Terms: conditions — Depression; Bipolar Disorder | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Quetiapine (Experimental): 18 patients of the risk-group will receive quetiapine (Seroquel Prolong (c)) for 8 weeks in adjunction to their antidepressant standard therapy. Group allocation is randomised and double-blind.
  Dosages: 50mg (day 1-3), 100mg (day 4-6) and 150mg (from day 7 onwards). Administration: Quetiapine will be given once daily before bedtime, not together with a meal and swallowed as a whole.
  Interventions: Drug: Quetiapine
- Placebo (Placebo Comparator): 18 patients of the risk-group will receive placebo for 8 weeks in adjunction to their antidepressant standard therapy. Group allocation is randomised and double-blind.
  The placebo does not contain any psychoactive substance.
  Interventions: Drug: Placebo
- Control-group (No Intervention): 18 depressive patients without a heightened risk for BPD will not receive any medication apart from their standard antidepressant therapy (control-group).

INTERVENTIONS:
Drug: Quetiapine — See information in arm description.
  Other Names: Seroquel Prolong
  Arms: Quetiapine
Drug: Placebo — See information in arm description.
  Arms: Placebo

SUMMARY:
Bipolar disorder (BPD) is often misdiagnosed as unipolar depression. This leads to inadequate treatment and can have negative impact on the course of the disease. There is now preliminary evidence that patients with unipolar and bipolar depression as well as healthy individuals with a heightened risk of BPD can be distinguished from each other based on their brain activity patterns and functional connectivity during resting state.

However, the impact of pharmacological treatment on these functional brain measures have not yet been clarified. For common antidepressants it has been shown that they seem to normalise aberrant brain activity patterns and functional connectivity. The problem is that some antidepressants can induce mania or accelerate pathological cycling in depressive patients with unrecognised BPD. Therefore, pharmacological drugs with mood-stabilising properties such as quetiapine are more and more prescribed. Although the effectiveness and tolerability have been proven, the neuronal effects of these adjunctive treatments are not clear. The aim of the study is thus to investigate the impact of quetiapine on measures of brain activity in depressive patients with a heightened risk of BPD. Moreover, the investigators want to examine whether the investigators can distinguish depressive patients with a heightened risk of BPD from depressive patients without a heightened risk of BPD using neuroimaging techniques, and whether these measures can predict the course of the disease.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of depressive episode (F32.X, F33.X) with duration less than < 6 months
* max. three previous episodes of illness
* no manic or hypomanic episodes in the past
* current treatment with one antidepressant
* MRI-compatibility
* unequivocal understanding of study information and autonomous consent
* for women: negative pregnancy test
* for risk-group:

  * 14 or more points on hypomania checklist (HCL-32)
  * additionally at least one of the following four risk factors:

    1. positive family history (i.e. first or second order relatives with BPD, schizoaffective or schizophrenic psychosis, mania or suicide attempt)
    2. initial manifestation before 30 years of age
    3. initial manifestation after childbirth
    4. suicide attempt in the past

Exclusion Criteria:

* additional diagnoses of psychiatric disorders (Organic, including symptomatic, mental disorders [F0X.X]; mental and behavioural disorders due to psychoactive substance use [F1X.X]; schizophrenia, schizotypal and delusional disorders [F2X.X]; mental retardation [F7X.X])
* chronic or acute physical disease
* individuals who are in a dependence- or work-relation with the sponsor
* limited or annulled legal capacity
* court or administrative order for hospitalisation
* for women: pregnancy, nursing period or unsafe contraceptive methods
* for the risk group:

  * clinical relevant changes in clinical chemistry, hematology, EEG or EKG
  * known contraindication for quetiapine (e.g. hypersensitivity to [active] ingredient[s], HIV-protease inhibitors, antimycotics, antibiotics)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
BOLD signal during a combined inhibition-reward-task | Baseline (Day 0)
  At baseline (day 0) the risk-group and control-group will be compared on BOLD signal (and behavioural data) during a combined inhibition-reward-task (neuronal correlate of cognitive control) (fMRI).
  These measures will be obtained once again at visit 4 (day 56) in the risk-group to evaluate the impact of quetiapine (i.e. change from baseline measure).
Functional connectivity in the default mode network during resting state (rstfMRI) | Baseline (Day 0)
  At baseline (day 0) the risk-group and control-group will be compared on functional connectivity in the default mode network during resting state (rstfMRI).
Structural differences in brain anatomy (MRI) | Baseline (Day 0)
  At baseline (day 0) the risk-group and control-group will be compared on structural differences in brain anatomy (MRI).
Structural integrity of nerve fibres (DTI) | Baseline (Day 0)
  At baseline (day 0) the risk-group and control-group will be compared on structural integrity of nerve fibres (DTI).
Effect of quetiapine on brain measures | Visit 4 (Day 56)
  After the quetiapine/ placebo intervention the risk-group will be compared whether there are changes from baseline in outcome measures 1 to 4.

SECONDARY OUTCOMES:
Plasma levels of quetiapine | Visit 4 (Day 56)
  Blood samples of the patients of the risk group will be obtained to analyse the plasma levels of quetiapine.
Change over time in affect and psychopathology | Baseline (Day 0), Visit 4 (Day 56), Follow-up (after 1 year)
  All patients (risk-group and control group) will be assessed with questionnaires tapping affect and psychopathology (MADRS, YMRS, CGI, PANSS, BDI-II, Bf-S, SWN-K, EPS, BARS, C-SSRS, NGASR). These measures will be obtained at three different time points to evaluate the respective change over time.
Personality | Baseline (Day 0)
  All patients (risk-group and control group) will be assessed with questionnaires of personality (TCI-R, BIS-15, RS-13).

CONTACTS AND LOCATIONS:
Overall Officials: Frank Schneider, Univ.-Prof., Study Director — University Hospital, Aachen
Locations (1):
- Clinic for psychiatry, psychotherapy and psychosomatic, RWTH Aachen University Hospital, Aachen, North Rhine-Westphalia, Germany